CLINICAL TRIAL: NCT06312956
Title: Multidimensional Evaluation of Patients' Affected by Obstructive Apnea Syndrome (OSAS) Before and After Ventilotherapy
Acronym: MULTI-OSAS
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C403
Record Dates: First submitted 2024-02-21; First posted 2024-03-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea; Sleep Disorder; Well-Being, Psychological; Cognitive Impairment; Cognitive Change; Neurologic Signs
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders; Psychological Well-Being; Cognitive Dysfunction; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for biomarkers analysis (i.e., orexin, histamine, light chain neurofilaments, Ab42, Ab40)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous Positive Airway Pressure Ventilotherapy — Breathing support device during sleeping
  Other Names: CPAP

SUMMARY:
This observational study aims to evaluate multiple dimensions of health in patients with Obstructive Sleep Apnea Syndrome (OSAS), before and after three weeks of ventilotherapy.

Specifically, the study aims to identify pre- vs post-treatment differences in the following domains:

* cognitive performance
* blood expression of biomarkers related to neurodegeneration
* psychosocial wellbeing

Thus, patients will complete the following evaluations before (T0) and after (T1) ventilotherapy:

* neuropsychological standard assessment
* blood sampling
* psychosocial self-reported questionnaires

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome is associated with cognitive difficulties, low psychosocial wellbeing and quality of life; however, the possible beneficial contribution of ventilotherapy on these dimensions is not completely clear. Ventilotherapy restores brain oxygenation and improve rest, possibly increasing cognitive performances, psychosocial health and quality of life. Multidisciplinary approaches to the treatment of OSAS are rare, although recommended. Solid proof of OSAS comorbidities may encourage clinicians to adopt a holistic perspective of care, leading to better rehabilitative outcomes. Also, evidence of the beneficial effects of ventilotherapy could increase patients' compliance to ventilotherapy, which is generally low.

The study aims to evaluate multiple dimensions of patient's health before and after three weeks of ventilotherapy, focusing on the cognitive performance, the blood expression of biomarkers related to neurodegeneration, and individual's psychosocial wellbeing.

Overall, it is expected improved cognitive performances and psychosocial wellbeing after ventilotherapy. Also, a reduction in the blood expression of biomarkers related to neurodegeneration (if found before the treatment) is hypothesized, although the limited research in this field requires cautious predictions.

Comprehensive evidence about OSAS comorbidity, beyond breath and sleep difficulties, is mandatory to design innovative multidisciplinary rehabilitative approaches in line with a holistic perspective of care. Effective multidisciplinary approaches are considered the gold standard in medical care, leading to better treatment outcomes and higher patients' satisfaction.

Beyond the clear ethical implication of providing higher quality of treatment, multidisciplinary interventions also imply a shared responsibility of treatment, preventing from clinical misjudgments and professionals' burnout.

ELIGIBILITY:
Inclusion Criteria:

* OSAS diagnosis (AHI > 5)
* handedness: right

Exclusion Criteria:

* previous ventilotherapy
* neurological and/or neurodegenerative conditions
* Personality disorders, autism spectrum disorders, schizophrenia, psychosis
* sleep disorders comorbidities (eg., narcolepsy)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individual affected by OSAS
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall cognitive functioning | baseline and after 3 weeks
  Montreal Cognitive Assessment MoCA (score range: 0-30; higher scores indicate higher cognitive functioning)
Selective attention | baseline and after 3 weeks
  Multiple Features Target Cancellation (MFTC) test (accuracy score range from 0 to 1; higher score suggest better performance)
Memory and learning | baseline and after 3 weeks
  Selective Reminding Test - SRT: three scores are provided. 1) long term memory storage capacity (0-72), learning (0-72), delayed recall (0-12). Higher scores indicate better performance.
Visuo-spatial abilities | baseline and after 3 weeks
  Rey Figure - copy: test score range from 0 to 36, higher scores indicate better performance
Inhibition | baseline and after 3 weeks
  Stroop Test: higher time scores and error scores indicate worst inhibitory control
Planning | baseline and after 3 weeks
  Tower of London - ToL: higher time score ( 0-36) and accuracy score (0-36) indicate better performance
Decision making | baseline and after 3 weeks
  Balloon Analog Risk Task - BART (test score)

SECONDARY OUTCOMES:
biomarkers of neurodegeneration | baseline and after 3 weeks
  blood concentration (pg/ml)
psychosocial wellbeing and satisfaction | baseline and after 3 weeks
  Psychological General Well-Being Index (i.e., test scores)
Quality of life (perceived psycho-physical and socio-economic wellbeing and satisfaction) | baseline and after 3 weeks
  Quality of Life Scale: 16-items self-report scored from 1 - terrible to 7 - delighted (score range 16-112); higher score indicate higher wellbeing and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano, Piancavallo, VCO, Italy

IPD SHARING:
Plan to Share IPD: No